CLINICAL TRIAL: NCT03243240
Title: Role of Triphasic Computed Tomography Imaging in the Detection of Acute Non-variceal Gastrointestinal Bleeding
Brief Title: Computed Tomography in Gastrointestinal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada abdelsabour, principle investigator, Assiut University
Other Study IDs: CT git bleeding
Record Dates: First submitted 2017-07-10; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: mutlidetector computed tomography — Multidetector computed tomography angiography with 16- MSCT scanner, medical system bright speed. Our protocol will include non-enhanced scanning then perform a triphasic angiography that includes arterial, portal and venous phases to detect acute gastrointestinal bleeding.
  Images will be acquired with the following parameters slice thickness 5mm for the unenhanced phase and 1.25mm for the arterial phase and porto-venous phases

SUMMARY:
Gastrointestinal bleeding represents a serious clinical problem and a common cause of hospitalisation with a mortality rate of 6-10% for upper Gastrointestinal bleeding and of 4% for lower Gastrointestinal bleeding requires a multidisciplinary approach involving gastroenterologists, endoscopists, surgeons and radiologists.

Gastrointestinal bleeding is self-limited in 80% of cases requiring only supportive measures. However, the persistence of bleeding represents a diagnostic challenge to locate the site of bleeding especially in severe bleeding and to determine, if possible its cause. This will allow to select the most appropriate therapeutic approach in order to reduce the morbidity and mortality, the length of hospitalisation and the transfusion requirements.

Current diagnostic algorithms vary widely from institution to institution and from clinician to clinician. Imaging modalities remain the mainstay of the diagnostic approach. They include endoscopy, video capsule, radionuclide imaging, catheter angiography and multidetector computed tomography imaging.

In recent years, Multidetector computed tomography has emerged as a promising technology to evaluate Gastrointestinal bleeding. The modality's ease of use and rapid results favour its use in any emergent situation. In addition, today's high-speed, narrow collimation multi-detector technology allows a large coverage area with minimal motion artifacts, with the ability to capture both arterial and venous phase with ease. Multidetector computed tomography is being increasingly used as this is a widely available, non-invasive and fast diagnostic technique that allows for visualisation of the entire intestinal tract and its lesions, the identification of vascularity and possible vascular abnormalities.

DETAILED DESCRIPTION:
A number of 30 Patients with Acute Gastrointestinal bleeding will be included in the study.

To maximise detection capabilities, it is crucial that Computed tomography angiography should begin as soon as possible while the patient is actively bleeding. Patients with active Gastrointestinal bleeding are assigned to intensive care units, and patients in shock are promptly resuscitated. Intensive care unit physicians provide appropriate monitoring for hemodynamically unstable patients undergoing Multidetector computed tomography angiography. Multidetector computed tomography angiography should be performed without prior oral administration of water or contrast material. Active contrast material extravasation within the bowel lumen is obscured by oral contrast material, leading to false-negative results.

Data acquisition: Investigators will perform Multidetector computed tomography angiography with 16- Multislice computed tomography scanner, medical system bright speed. The protocol will include non-enhanced scanning then perform a triphasic angiography that includes arterial, portal and venous phases to detect acute Gastrointestinal bleeding.

Images will be acquired with the following parameters slice thickness 5mm for the unenhanced phase and 1.25mm for the arterial phase and Porto-venous phases, pitch 1.375, 300 Miliambiar, 120kilovolt and rotation time 0.7 seconds.

Images acquired are reconstructed for coronal, sagittal, Volume Rendering and Maximum Intensity Projection images. A similar protocol may be used with a 64-Multislice computed tomography scanner.

A dose of 1-2 ml/kg body weight of concentration 370mg/ml non-ionized contrast media will be administered at a rate of 4ml/sec, with an upper limit of 150ml. Venous access is an antecubital vein with a 14 or at least 18G cannula. The scan delay time for the arterial phase images is obtained by using bolus tracking with a circular region of interest positioned in the abdominal aorta and a predefined 90-housenfield unit bolus-trigger threshold to the start of automatic scanning. The coverage from just above the diaphragm to the Ischial tuberosities including the rectum in all cases.

Study interpretation post processing will be performed with a 4.6 version workstation. All studies are reviewed in the axial plane and with multiplanar reformation images. Real-time maximum-intensity projection images facilitate rapid study interpretation for optimal case management.

The radiologist will try to get the following information:

* presence or absence of bleeding.
* localise the site of bleeding.
* detect the cause of bleeding: tumour, Arteriovenous malformations….. The confirmation of the triphasic Multislice computed tomography results will be done by angiographic intervention and embolization of bleeding vessel

ELIGIBILITY:
Inclusion Criteria:

* patients with unexplained non variceal gastrointestinal bleeding

Exclusion Criteria:

* patients with impaired renal functions or terminal liver failure. pregnancy. patients known to be sensitive to contrast media. cases diagnosed endoscopically as variceal bleeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A number of 30 Patients with Acute Gastrointestinal bleeding will be included in the study.
  This study will be performed in Radio diagnostic department in Assiut University Hospital.
  We will perform multi detector computed tomography angiography with 16 or 64 multi slice computed tomography scanner.
  our protocol will include non enhanced scanning then perform triphasic angiography that include arterial , portal and venous phases to detect gastrointestinal bleeding.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Role of triphasic computed tomography imaging in detection of acute non variceal gastrointestinal tract bleeding | one year
  Number of 30 patients with acute gastrointestinal bleeding will undergo multislice computed tomography angiography with 16 multislice computed tomography scanner with dose 1-2ml/kg body weight contrast media and the study will be revised to detect the contrast extravasation which means active bleeding, and will detect the cause of bleeding such as tumor, aneurysm, arteriovenous malformation....and confirmation of these results will be done by angiographic intervention and embolization of the bleeding vessel

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abdelsabour, resident, Principal Investigator — Assiut University

REFERENCES:
- [Background] Geffroy Y, Rodallec MH, Boulay-Coletta I, Julles MC, Ridereau-Zins C, Zins M. Multidetector CT angiography in acute gastrointestinal bleeding: why, when, and how. Radiographics. 2011 May-Jun;31(3):E35-46. doi: 10.1148/rg.313105206. PMID 21721196